CLINICAL TRIAL: NCT01582269
Title: A Phase 2 Study of LY2157299 Monohydrate Monotherapy or LY2157299 Monohydrate Plus Lomustine Therapy Compared to Lomustine Monotherapy in Patients With Recurrent Glioblastoma
Brief Title: A Study in Recurrent Glioblastoma (GB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13849; H9H-MC-JBAL (Other: Eli Lilly and Company); 2011-004418-40 (EudraCT Number)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — LY-2157299; Lomustine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Galunisertib (Experimental): * Participants received Galunisertib 300 milligrams (mg) orally twice daily (BID) for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Treatment continued until disease progression, death, or discontinuation criteria were met.
  Interventions: Drug: Galunisertib
- Arm B: Galunisertib + Lomustine (Experimental): * Participants received Galunisertib 300 mg orally BID for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Participants received a first dose of Lomustine at 100 milligrams per square meter (mg/m²) administered orally. Thereafter, starting with the second dose, Lomustine was administered orally once every 6 weeks at 100-130 mg/m², at the discretion of the investigator.
  * Treatment continued until disease progression, death, or discontinuation criteria were met.
  Interventions: Drug: Galunisertib; Drug: Lomustine
- Arm C: Lomustine + Placebo (Active Comparator): * Participants received a first dose of Lomustine at 100 mg/m² administered orally. Thereafter, starting with the second dose, Lomustine was administered orally once every 6 weeks at 100-130 mg/m², at the discretion of the investigator.
  * Participants received Galunisertib-matched Placebo orally BID for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Treatment continued until disease progression, death, or discontinuation criteria were met.
  Interventions: Drug: Lomustine; Drug: Placebo

INTERVENTIONS:
Drug: Galunisertib — Administered orally
  Other Names: LY2157299 monohydrate
  Arms: Arm A: Galunisertib; Arm B: Galunisertib + Lomustine
Drug: Lomustine — Administered orally
  Arms: Arm B: Galunisertib + Lomustine; Arm C: Lomustine + Placebo
Drug: Placebo — Administered orally
  Other Names: Galunisertib-matched Placebo
  Arms: Arm C: Lomustine + Placebo

SUMMARY:
The purpose of the study is to see whether treatment with LY2157299 on its own, LY2157299 plus lomustine therapy or lomustine plus placebo can help participants with brain cancer

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed diagnosis of relapsed intracranial GB
* Progressive Disease (PD) following standard chemoradiation
* Prior surgical resection allowed
* Performance status Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Adequate hematologic, hepatic and renal function
* Discontinued all prior cancer treatments for cancer & recovered from the acute effects of therapy
* Tumor specimen must be available for a central pathology review and prognostic and predictive biomarker evaluation

Exclusion Criteria:

* Moderate or severe heart disease based on New York Heart Association (NYHA) criteria
* Prior nitrosurea therapy (including lomustine or Gliadel)
* Prior bevacizumab as 1st line treatment for GB (if treatment was concluded 12 months prior to enrollment, the patient may be eligible to participate in the trial)
* Current acute or chronic myelogenous leukemia
* Second primary malignancy that may affect the interpretation of results
* Serious concomitant systemic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-04-26 (Actual); Primary Completion 2014-07-26 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bobigny
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nancy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz, Poland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona, Spain

REFERENCES:
- [Derived] Smith CL, Thomas Z, Enas N, Thorn K, Lahn M, Benhadji K, Cleverly A. Leveraging historical data into oncology development programs: Two case studies of phase 2 Bayesian augmented control trial designs. Pharm Stat. 2020 May;19(3):276-290. doi: 10.1002/pst.1990. Epub 2020 Jan 5. PMID 31903699
- [Derived] Brandes AA, Carpentier AF, Kesari S, Sepulveda-Sanchez JM, Wheeler HR, Chinot O, Cher L, Steinbach JP, Capper D, Specenier P, Rodon J, Cleverly A, Smith C, Gueorguieva I, Miles C, Guba SC, Desaiah D, Lahn MM, Wick W. A Phase II randomized study of galunisertib monotherapy or galunisertib plus lomustine compared with lomustine monotherapy in patients with recurrent glioblastoma. Neuro Oncol. 2016 Aug;18(8):1146-56. doi: 10.1093/neuonc/now009. Epub 2016 Feb 21. PMID 26902851

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All the treated participants who experienced progressive disease or died were considered study completers, while those who withdrew consent or were lost to follow-up were not.
Groups:
- Arm A: Galunisertib: * Participants received Galunisertib 300 milligrams (mg) orally twice daily (BID) for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Treatment continued until disease progression or discontinuation criteria were met.
- Arm B: Galunisertib + Lomustine: * Participants received Galunisertib 300 mg orally BID for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Participants received a first dose of Lomustine at 100 milligrams per square meter (mg/m²) administered orally. Thereafter, starting with the second dose, Lomustine was administered orally once every 6 weeks at 100-130 mg/m², at the discretion of the investigator.
  * Treatment continued until disease progression or discontinuation criteria were met.
- Arm C: Lomustine + Placebo: * Participants received a first dose of Lomustine at 100 mg/m² administered orally. Thereafter, starting with the second dose, Lomustine was administered orally once every 6 weeks at 100-130 mg/m², at the discretion of the investigator.
  * Participants received Galunisertib-matched Placebo orally BID for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Treatment continued until disease progression or discontinuation criteria were met.
Period: Overall Study
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo
Started | 39 | 79 | 40
Received at Least One Dose of Study Drug | 39 | 79 | 40
Safety Analysis Population (All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received.) | 40 | 78 (One female participant assigned to Arm B received only Galunisertib monotherapy (i.e., did not receive Lomustine). Therefore, for safety analysis that participant was excluded from arm B and counted under Arm A, Thus, Arm A = 40 and Arm B=78.) | 40 (One participant assigned to Arm C received only Placebo (i.e., did not receive Lomustine) and was therefore reported separately for safety analyses based on actual treatment received Arm C: Lomustine + Placebo = 39; Arm C: Lomustine + Placebo (Placebo Alone) = 1.)
Completed | 38 | 79 | 40
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Arm A: Galunisertib: * Participants received Galunisertib 300 mg orally BID for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Treatment continued until disease progression, death, or discontinuation criteria were met.
- Arm B: Galunisertib + Lomustine: * Participants received Galunisertib 300 mg orally BID for 14 days, followed by 14 days of rest in a 28-day cycle.
  * Participants received a first dose of Lomustine at 100 mg/m² administered orally. Thereafter, starting with the second dose, Lomustine was administered orally once every 6 weeks at 100-130 mg/m², at the discretion of the investigator.
  * Treatment continued until disease progression, death, or discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo | Total
Number analyzed (Participants) | 39 | 79 | 40 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.9) | 57.5 (9.3) | 56.9 (10.2) | 57.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 17 | 56
  Male | 21 | 58 | 23 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 2 | 11
  Not Hispanic or Latino | 29 | 56 | 27 | 112
  Unknown or Not Reported | 7 | 17 | 11 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 30 | 60 | 29 | 119
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 16 | 10 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 3 | 1 | 4
  Belgium | 3 | 8 | 3 | 14
  United States | 7 | 8 | 6 | 21
  Poland | 1 | 1 | 0 | 2
  Italy | 8 | 14 | 8 | 30
  Australia | 4 | 14 | 2 | 20
  France | 7 | 17 | 11 | 35
  Germany | 4 | 7 | 5 | 16
  Spain | 5 | 6 | 3 | 14
  Netherlands | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until death from any cause. For participants not known to have died by the data-inclusion cutoff date, OS is censored at the last date they were known to be alive.
Time Frame: Randomization to Date of Death from Any Cause (Up To 20.5 Months)
Population: All randomized participants who received at least one dose of study drug (including the censored participants). Number of participants censored in Arm A: Galunisertib = 9; Arm B: Galunisertib + Lomustine = 8; and Arm C: Lomustine + Placebo = 6.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo
Number analyzed (Participants) | 39 | 79 | 40
Months | 8.0 [NA to NA] — 95% credible interval (5.7 to 11.7) | 6.7 [NA to NA] — 95% credible interval (5.3 to 8.5) | 7.5 [NA to NA] — 95% credible interval (5.6 to 10.3)
Statistical Analysis 1: Comparison: Arm A: Galunisertib vs Arm C: Lomustine + Placebo; The Bayesian analyses below include credible intervals rather than confidence intervals for the hazard ratios; Test type: Superiority; Bayesian exponential-likelihood model; Hazard Ratio (HR) = 0.9336, 95% CI 2-sided [0.58 to 1.49]; The posterior probability treatment difference is 0.6158
Statistical Analysis 2: Comparison: Arm B: Galunisertib + Lomustine vs Arm C: Lomustine + Placebo; The Bayesian analyses below include credible intervals rather than confidence intervals for the hazard ratios; Test type: Superiority; Bayesian exponential-likelihood model; Hazard Ratio (HR) = 1.1290, 95% CI 2-sided [0.78 to 1.65]; The posterior probability treatment difference is 0.2628

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of the first observation of objective disease progression or death from any cause, whichever occurred first. Participants known to be alive and without disease progression were censored at the date of their last objective progression-free disease assessment prior to the initiation of any subsequent systemic anticancer therapy.
Time Frame: Randomization to Objective Progression or Death Due to Any Cause (Up To 19 Months)
Population: All randomized participants who received at least one dose of study drug (including the censored participants). Number of participants censored in Arm A: Galunisertib = 7; Arm B: Galunisertib + Lomustine = 8; and Arm C: Lomustine + Placebo = 4.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo
Number analyzed (Participants) | 39 | 79 | 40
Months | 1.8 [1.6 to 3.0] | 1.8 [1.7 to 1.8] | 1.9 [1.7 to 1.9]

3. Secondary Outcome: Percentage of Participants With Tumour Response
Description: Tumour response was assessed using Response Assessment in Neuro-Oncology (RANO) criteria. Responses included Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD). CR required disappearance of all enhancing lesions, no new lesions, stable or improved non-enhancing lesions, and no corticosteroid use. PR was defined as ≥50% reduction in enhancing lesion size, no new lesions, stable or improved non-enhancing lesions, and stable or reduced corticosteroid use. SD indicated no significant change in lesion size or clinical status. PD was defined as ≥25% increase in lesion size, new lesions, or clinical deterioration. Percentage of participants with tumor response is defined as the percentage of participants who achieved these tumor responses based on RANO criteria.Participants whose tumor response could not be assessed due to inadequate imaging data were categorized as 'Unknown'.
Time Frame: Randomization until measured progressive disease (Up To 19 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo
Number analyzed (Participants) | 39 | 79 | 40
Percentage of participants
  CR | 0.0 | 1.3 | 0.0
  PR | 5.1 | 0.0 | 0.0
  SD | 25.6 | 20.3 | 30.0
  PD | 53.8 | 63.3 | 65.0
  Unknown | 15.4 | 15.2 | 5.0

4. Secondary Outcome: Population Pharmacokinetics (PopPK): Absorption Rate Constant of Galunisertib (Arm A: Galunisertib and Arm B: Galunisertib + Lomustine)
Description: The absorption rate constant (Ka) of Galunisertib was estimated using PopPK modeling based on plasma concentration-time data collected during Cycle 1. A two-compartment model with first-order absorption was applied using nonlinear mixed-effects modeling. Samples were collected at the following time points: Cycle 1 Day 1: Predose, 0.5-2 hours (h), 3.5-5 h, and 48 h post-dose; Day 14: Predose, 0.5-2 h, 3.5-5 h, 24 h, and 48 h post last dose. Individual participant Ka values were derived from model-estimated parameters using all available PK timepoints.The reported outcome is the mean of these individual Ka estimates across both treatment arms (Arm A: Galunisertib; Arm B: Galunisertib + Lomustine).
Time Frame: Cycle (C) 1: Day (D)1: Predose, 0.5-2 hours (h), 3.5-5 h, and 48 h post-dose; Day 14: Predose, 0.5-2 h, 3.5-5 h, 24 h, and 48 h post last dose
Population: All randomized participants who received at least one dose of Galunisertib (Arm A and Arm B) and had evaluable PK data were included in the analysis. As prespecified in the statistical analysis plan, PK analyses of Galunisertib exposure parameters were conducted using data combined from both arms.
Measure: Mean (Standard Error); unit: One per hour (1/hour)
Groups:
- Arm A: Galunisertib and Arm B: Galunisertib + Lomustine: * Arm A: Galunisertib: Participants received Galunisertib 300 mg orally BID for 14 days, followed by 14 days of rest in a 28-day cycle until disease progression, death, or discontinuation criteria were met.
  * Arm B: Galunisertib + Lomustine: Participants received Galunisertib 300 mg orally BID for 14 days, followed by 14 days of rest in a 28-day cycle, plus received a first dose of Lomustine at 100 mg/m² administered orally. Thereafter, starting with the second dose, Lomustine was administered orally once every 6 weeks at 100-130 mg/m², at the discretion of the investigator, until disease progression, death, or discontinuation criteria were met.
Arm/Group | Arm A: Galunisertib and Arm B: Galunisertib + Lomustine
Number analyzed (Participants) | 114
One per hour (1/hour) | 2.28 (26)

5. Secondary Outcome: Population Pharmacokinetics (PopPK): Mean Steady State Apparent Volume of Distribution (Vss) of Galunisertib (Arm A: Galunisertib and Arm B: Galunisertib + Lomustine)
Description: The Vss at steady state of Galunisertib was estimated using PopPK modeling based on plasma concentration-time data collected during Cycle 1.A two-compartment model was applied using nonlinear mixed-effects modeling. Samples were collected at the following time points: Cycle 1 Day 1: Predose, 0.5-2 hours (h), 3.5-5 h, and 48 h post-dose; Day 14: Predose, 0.5-2 h, 3.5-5 h, 24 h, and 48 h post last dose. Individual participant Vss values were derived from model-estimated parameters using all available PK timepoints. The reported outcome is the mean of individual Vss estimates across both treatment arms (Arm A: Galunisertib; Arm B: Galunisertib + Lomustine).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Liters (L)
Arm/Group | Arm A: Galunisertib and Arm B: Galunisertib + Lomustine
Number analyzed (Participants) | 114
Liters (L) | 175 (8.9)

6. Secondary Outcome: Population Pharmacokinetics (PopPK): Mean Population Clearance of Galunisertib (Arm A: Galunisertib and Arm B: Galunisertib + Lomustine)
Description: The apparent clearance (CL/F) of Galunisertib was estimated using PopPK modeling based on plasma concentration-time data collected during Cycle 1. A two-compartment model was applied using nonlinear mixed-effects modeling. Samples were collected at the following time points: Cycle 1 Day 1: Predose, 0.5-2 hours (h), 3.5-5 h, and 48 h post-dose; Day 14: Predose, 0.5-2 h, 3.5-5 h, 24 h, and 48 h post last dose. Individual participant CL/F values were derived from model-estimated parameters using all available PK timepoints. The reported outcome is the mean of these individual CL/F estimates across both treatment arms (Arm A: Galunisertib; Arm B: Galunisertib + Lomustine).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Liter per hour (L/hr)
Arm/Group | Arm A: Galunisertib and Arm B: Galunisertib + Lomustine
Number analyzed (Participants) | 114
Liter per hour (L/hr) | 37.5 (5.0)

7. Secondary Outcome: Change From Baseline in Neurocognitive Function Using Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: The Hopkins Verbal Learning Test-Revised comprises:
  * 3 Learning Trials: Participants were presented with a list of 12 words (from 3 semantic categories) and were asked to recall them to test verbal learning and memory.
  * Delayed Recall Trial: Conducted 20-25 minutes after the 3rd learning trial to test memory retention.
  * Delayed Recognition Trial: Participants identified previously presented words from a list that included 12 distractors to test recognition discrimination.
  Scoring Components:
  * Total Recall Score (0-36): Sum of correctly recalled words across the 3 learning trials.
  * Delayed Recall Score (0-12): Number of correct words recalled after the delay.
  * Recognition Discrimination Index Score (+12 to -12): Calculated as the number of true positives (correctly identified words) minus false positives (incorrectly identified words, i.e., distractors).
  For each of the 3 reported scores, higher scores = better neurocognitive performance; lower scores = decline.
Time Frame: Baseline, Month 20
Population: All randomized participants who received at least one dose of the study drug and had a baseline and at least one post-baseline measurement for this outcome.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo
Number analyzed (Participants) | 36 | 74 | 39
Score on a scale
  Total Recall Score | -0.2 (1.4) | -0.2 (1.2) | -0.3 (1.5)
  Delayed Recall Score: number analyzed (Participants) | 35 | 71 | 39
  Delayed Recall Score | -0.8 (2.2) | 0.0 (1.4) | 0.1 (1.3)
  Recognition Discrimination Index Score: number analyzed (Participants) | 35 | 71 | 39
  Recognition Discrimination Index Score | -1.3 (5.1) | 0.7 (4.1) | 0.1 (2.0)

8. Secondary Outcome: Change From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom and Interference Severity Scores: (Brain Tumor Symptoms, Core Symptoms, Interference Symptoms)
Description: The MDASI-BT assesses the severity of multiple brain tumor-related symptoms and the impact of these symptoms on daily functioning in the last 24 hours. It includes:
  * 13 core symptoms measuring severity of pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, memory problems, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness/tingling, rated 0-10, where 0 = "not present" and 10 = "as bad as you can imagine."
  * 9 brain tumor-specific symptoms assess severity of difficulty speaking, weakness, seizures, difficulty understanding, vision changes, appearance changes, bowel pattern changes, concentration problems, and irritability, rated 0-10, where 0 = "not present" and 10 = "as bad as you can imagine."
  * 6 interference items assess impact on general activity, mood, work, relations, walking, and enjoyment of life, rated 0-10, where 0 = "did not interfere" and 10 = "interfered completely."
Time Frame: Baseline, Month 21
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo
Number analyzed (Participants) | 38 | 77 | 38
Score on a scale
  Brain Tumor Symptoms | 0.0 (2.3) | 0.3 (1.9) | -0.3 (1.9)
  Core Symptoms | 0.0 (1.5) | 0.3 (1.5) | 0.3 (0.9)
  Interference Symptoms: number analyzed (Participants) | 37 | 77 | 38
  Interference Symptoms | 0.2 (2.8) | 0.8 (2.2) | 1.1 (3.0)

ADVERSE EVENTS:
Time Frame: Baseline Up to 11 years 4 months
Description: * Adverse events were reported for the "Safety Analysis Population."
  * Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Arm C: Lomustine + Placebo (Placebo Alone): • Participants randomized to Arm C who did not receive the planned treatment but received Galunisertib-matched placebo alone were categorized under this group.
Arm/Group | Arm A: Galunisertib | Arm B: Galunisertib + Lomustine | Arm C: Lomustine + Placebo | Arm C: Lomustine + Placebo (Placebo Alone)
All-Cause Mortality (participants affected / at risk) | 37/40 | 75/78 | 38/39 | 1/1
Serious Adverse Events (participants affected / at risk) | 21/40 | 31/78 | 15/39 | 1/1
Other Adverse Events (participants affected / at risk) | 34/40 | 69/78 | 31/39 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Galunisertib (N=40) | Arm B: Galunisertib + Lomustine (N=78) | Arm C: Lomustine + Placebo (N=39) | Arm C: Lomustine + Placebo (Placebo Alone) (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eastern cooperative oncology group performance status worsened (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 3 (3) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Iiird nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-24-hour sleep-wake disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 7 (8) | 4 (4) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A: Galunisertib (N=40) | Arm B: Galunisertib + Lomustine (N=78) | Arm C: Lomustine + Placebo (N=39) | Arm C: Lomustine + Placebo (Placebo Alone) (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 4 (5) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 9 (11) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (10) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 21 (26) | 12 (12) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (7) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 7 (9) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 5 (8) | 6 (7) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 13 (13) | 8 (10) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 14 (16) | 8 (11) | 0 (0)
Asthenia (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (10) | 20 (25) | 14 (15) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (6) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (7) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (12) | 3 (4) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 4 (5) | 4 (4) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 6 (9) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 3 (3) | 5 (5) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 6 (13) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (15) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (7) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 3 (3) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 6 (7) | 4 (4) | 3 (3) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 8 (9) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 20 (27) | 10 (13) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 7 (9) | 6 (6) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 5 (5) | 4 (6) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 6 (7) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (3) | 5 (5) | 5 (5) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 3 (4) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/19 (1) | 0/20 (0) | 0/17 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (11) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (7) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1/19 (1) | 0/20 (0) | 0/17 (0) | 0/0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT01582269/Prot_000.pdf
  • Statistical Analysis Plan (2012-04-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT01582269/SAP_001.pdf